CLINICAL TRIAL: NCT03921294
Title: Prospective, Single-arm, Open-label Use of Hemlibra (Emicizumab) to Treat Hemophilic Pseudotumor
Brief Title: HemLibra Prophylaxis in Patients With Hemophilic Pseudotumor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Global COVID-19 pandemic prevented further study visits or enrollment.
Sponsor: Indiana Hemophilia &Thrombosis Center, Inc. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Amy D Shapiro, MD, Medical Director, Indiana Hemophilia &Thrombosis Center, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO-IIS-2018-10581
Record Dates: First submitted 2019-03-29; First posted 2019-04-19 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Haemophilic Pseudotumour
MeSH Terms: interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: single arm prospective open-label single-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients with hemophilic pseudotumor will be treated with prophylactic emicizumab and assessed for improvement.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — bispecific monoclonal antibody binding to activated Factor IX and Factor X
  Other Names: HemLibra

SUMMARY:
This is a single arm, phase 4, prospective, open-label, United States single-center study to assess the hemostatic efficacy and safety of Hemlibra (emicizumab) for hemostatic control of hemophilia A patients (baseline FVIII level <40%) with and without inhibitors with hemophilic pseudotumors; secondary outcomes will assess changes in quality of life and activity level in treated patients.

DETAILED DESCRIPTION:
This is a single arm, phase 4, prospective, open-label, United States single-center study to assess the hemostatic efficacy and safety of Hemlibra (emicizumab) for hemostatic control of hemophilia A patients, (baseline FVIII level <40%), children and adults, with and without inhibitors with hemophilic pseudotumors; secondary outcomes will assess changes in quality of life and activity level in treated patients.

Hemlibra (emicizumab) will be administered as primary weekly prophylaxis after the enrollment/screening visit is complete (approximately 7-10 days after screening, if laboratory results are available and eligibility is confirmed). If an activity monitoring device is typically utilized by the patient (eg, a Fitbit) then permission will be requested from the patient at screening to access the data for 1 month prior to screening as a baseline comparator for post-treatment activity. The use of an activity-monitoring device is not required by the study.

The enrollment period is 2 years and the study will last a maximum of 4 years; subjects will receive study medication (Hemlibra, emicizumab) for a minimum of 2 years and a maximum of 4 years based upon time of enrollment. Hemlibra (emicizumab) will be administered using the FDA-approved once-weekly dosing regimen for loading dose and prophylactic dose. Breakthrough bleeding events will be recorded and treated with locally available FVIII (eg, pdFVIII or rFVIII) in non-inhibitor subjects and inhibitor subjects with low titer inhibitors (titer<5 BU). The lowest dose of FVIII expected to achieve hemostasis will be utilized for treatment of breakthrough bleeding events in non-inhibitor and low-titer inhibitor patients. Subjects with high-titer inhibitors (titer ≥5 BU) and those with low titer inhibitors who do not respond to FVIII will be required to utilize rFVIIa as first line therapy; aPCC (<100 U/kg/day for preferably no more than 1 day) may only be used upon approval of the Study Investigator and under the supervision of a physician.

The proposed study is seeking to address the following knowledge gaps:

Does weekly prophylactic Hemlibra (emicizumab) reduce the rate of bleeding events in subjects with hemophilia A and pseudotumor, including the rate of hospitalization, anemia and transfusion? Does weekly prophylactic Hemlibra (emicizumab) control the progression of hemophilic pseudotumor? Does weekly prophylactic Hemlibra (emicizumab) result in an increase in QoL and activity level?

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form from the subject, parent or guardian
* Diagnosis of congenital hemophilia A (baseline FVIII level <40%) with or without FVIII inhibitor, either high or low responding, regardless of titer
* Diagnosis of a hemophilic pseudotumor confirmed by radiologic assessment such as CT or MRI
* Any weight or BMI
* Medical documentation of prophylactic or episodic treatment (FVIII or bypassing agent) and the number of bleeding episodes for at least 16 weeks, and up to 6 months if available, prior to entry into the study
* Medical documentation of any need for PRBC transfusion or hospitalization for 6 months prior to entry into the study
* Subjects with a history of an inhibitor should provide documentation of the inhibitor history including date of initial diagnosis of inhibitor, peak titer, and agent utilized for hemostatic control
* Subjects with high titer inhibitors or those with low titer inhibitors who do not respond to FVIII must be willing to use rFVIIa as first line therapy for the treatment of breakthrough bleeding events
* Medical documentation of ITI therapy for subjects with a history of a FVIII inhibitor and ITI, including current FVIII inhibitor titer
* Willingness to discontinue any current prophylactic hemostatic regimen (FVIII or bypassing agent) and/or FVIII ITI therapy for the duration of the study

  * Subjects receiving FVIII prophylaxis must be willing to discontinue their FVIII prophylactic regimen immediately prior to their second loading dose of Hemlibra (emicizumab)
  * Subjects receiving bypassing agent prophylaxis must be willing to discontinue their prophylactic regimen at least 24 hours prior to their first loading dose of Hemlibra (emicizumab)
  * Subjects receiving FVIII ITI therapy must be willing to discontinue ITI immediately prior to their first loading dose of Hemlibra (emicizumab)
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including the health-related questionnaires, activity tracking, and bleed diaries, using systems provided during the study
* Adequate hepatic function, defined as total bilirubin ≤1.5 × age-adapted upper limit of normal (ULN) (excluding Gilbert's syndrome) and both AST and ALT ≤3 × age-adapted ULN at the time of screening, and no clinical signs or known laboratory/radiographic evidence consistent with cirrhosis
* Subjects must be willing to be vaccinated against HAV and HBV if not previously vaccinated, exposed or immune to HAV or HBV*
* Adequate hematologic function, defined as a platelet count ≥100,000/μL and a PT≤1.5 times the ULN at the time of screening
* Adequate renal function, defined as serum creatinine ≤2.5 × age-adapted ULN and creatinine clearance ≥30 mL/min by Cockcroft-Gault formula
* For women with hemophilia of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 5 elimination half-lives (24 weeks) after the last dose of study drug

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than congenital hemophilia A
* Lack of a documented diagnosis of hemophilic pseudotumor
* Patients who are at high risk for TMA (eg, have a previous medical or family history of TMA), in the Study Investigator's judgment
* History of illicit drug or alcohol abuse within 48 weeks prior to screening, in the Study Investigator's judgment
* Previous (within the last 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Other conditions (eg, certain autoimmune diseases) that may currently increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the Emicizumab injection
* Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the study
* Known HIV infection with CD4 counts <200 cells/μL. HIV infection with CD4 counts ≥200 cells/μL permitted
* Use of systemic immunomodulators (eg, interferon) at enrollment or planned use during the study, with the exception of anti-retroviral therapy
* Concomitant disease, condition, significant abnormality on screening evaluations or laboratory tests, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the Study Investigator, pose an additional unacceptable risk in administering study drug to the patient
* Receipt of any of the following:

  * Hemlibra (emicizumab) in a prior investigational study
  * An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration
  * A non-hemophilia-related investigational drug within last 30 days or 5 half-lives, whichever is shorter
  * Any other investigational drug currently being administered or planned to be administered
* Inability to comply with the study protocol in the opinion of the Study Investigator
* Pregnancy or lactation or intention to become pregnant during the study
* Women with a positive serum pregnancy test result within 10 days prior to initiation of study drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Shapiro, MD, Principal Investigator — Indiana Hemophilia &Thrombosis Center, Inc.
Locations (1):
- Indiana Hemophila @Thrombosis Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share resources and data from this project through collaborative publications in the scientific literature as well as through national, regional and international conference presentations. We will also share our methods and findings in a prompt manner with regional, national and international stakeholders to ensure that findings will be readily available to other researchers and clinicians with clinical or scientific interest in the subject area. Individual participant data that underlie the results reports in publications, reports or presentations (including text, tables, figures and appendices) will be shared after de-identification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and additional information on study methods will be made available starting 9 months after publication or conclusion of the study and ending 36 months following publication or study conclusion.
Access Criteria: IPD and study information will be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary"), whose proposals are methodologically sound, and for purposes that are consistent with the aims of the underlying research. Proposals will be reviewed by the Principle Investigator, Dr. Amy Shapiro, and may be submitted to ashapiro@ihtc.org. Requestors will be required to sign a data access and use agreement.

REFERENCES:
- [Result] Ahlberg AK. On the natural history of hemophilic pseudotumor. J Bone Joint Surg Am. 1975 Dec;57(8):1133-6. PMID 1202003
- [Result] Blanchette VS, Key NS, Ljung LR, Manco-Johnson MJ, van den Berg HM, Srivastava A; Subcommittee on Factor VIII, Factor IX and Rare Coagulation Disorders of the Scientific and Standardization Committee of the International Society on Thrombosis and Hemostasis. Definitions in hemophilia: communication from the SSC of the ISTH. J Thromb Haemost. 2014 Nov;12(11):1935-9. doi: 10.1111/jth.12672. Epub 2014 Sep 3. No abstract available. PMID 25059285
- [Result] Franchini M, Mannucci PM. Hemophilia A in the third millennium. Blood Rev. 2013 Jul;27(4):179-84. doi: 10.1016/j.blre.2013.06.002. Epub 2013 Jun 28. PMID 23815950
- [Result] Gringeri A, Leissinger C, Cortesi PA, Jo H, Fusco F, Riva S, Antmen B, Berntorp E, Biasoli C, Carpenter S, Kavakli K, Morfini M, Negrier C, Rocino A, Schramm W, Windyga J, Zulfikar B, Mantovani LG. Health-related quality of life in patients with haemophilia and inhibitors on prophylaxis with anti-inhibitor complex concentrate: results from the Pro-FEIBA study. Haemophilia. 2013 Sep;19(5):736-43. doi: 10.1111/hae.12178. Epub 2013 Jun 4. PMID 23731246
- [Result] Liu SS, White WL, Johnson PC, Gauntt C. Hemophilic pseudotumor of the spinal canal. Case report. J Neurosurg. 1988 Oct;69(4):624-7. doi: 10.3171/jns.1988.69.4.0624. PMID 3418398
- [Result] Magallon M, Monteagudo J, Altisent C, Ibanez A, Rodriguez-Perez A, Riba J, Tusell J, Martin-Villar J. Hemophilic pseudotumor: multicenter experience over a 25-year period. Am J Hematol. 1994 Feb;45(2):103-8. doi: 10.1002/ajh.2830450202. PMID 8141115
- [Result] Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47. doi: 10.1111/j.1365-2516.2012.02909.x. Epub 2012 Jul 6. PMID 22776238
- [Result] van Ommeren JW, Mooren DW, Veth RP, Novakova IR, van de Kaa CA. Pseudotumor occurring in hemophilia. Arch Orthop Trauma Surg. 2000;120(7-8):476-8. doi: 10.1007/s004029900087. PMID 10968546
- See also: What is Hemophilia? — https://www.nhlbi.nih.gov/health/health-topics/topics/hemophilia/
- See also: WFH Guidelines for the management of hemophilia — http://www1.wfh.org/publication/files/pdf-1472.pdf
- See also: WFH report on the annual global survey 2011 — http://www1.wfh.org/publication/files/pdf-1488.pdf
- See also: WFH report on the annual global survey 2013 — http://www1.wfh.org/publications/files/pdf-1591.pdf
- See also: WFH report on the annual global survey 2015 — http://www1.wfh.org/publication/files/pdf-1669.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Emicizumab (Single Arm): Patients with hemophilic pseudotumor will be treated with prophylactic emicizumab and assessed for improvement. Emicizumab: bispecific monoclonal antibody binding to activated Factor IX and Factor X
Period: Overall Study
Arm/Group | Emicizumab (Single Arm)
Started | 1
Enrolled | 1
Completed Treatment | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with Factor VIII deficiency and hemophilia pseudotumor.
Groups:
- Baseline Characteristics: Patients with factor VIII deficiency and a hemophilic pseudotumor.
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 31 [31 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Hemostatic Efficacy of Prophylactic Weekly Injections of Hemlibra (Emicizumab) Based on Hemoglobin
Description: Maintenance or increase of hemoglobin (g/dl) from participants' baseline level based on serial blood tests.
Time Frame: Every 6 months, for the 2 years and 10 months of the patient's study participation duration.
Measure: Mean (Full Range); unit: gm/dL
Arm/Group | Single Arm
Number analyzed (Participants) | 1
gm/dL | 9.5 [8 to 11]

2. Primary Outcome: Hemostatic Efficacy of Prophylactic Weekly Injections of Hemlibra (Emicizumab) Based on Participants' Need for Blood Transfusions or Lack of
Description: Whether or not the patient requires blood transfusions (units of RBCs) due to blood loss secondary to lack of hemostatic efficacy during the duration of study treatment duration.
Time Frame: Every 6 months, for the 2 years and 10 months of the patient's study participation duration.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab (Single Arm)
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Breakthrough Bleeds
Description: Number of breakthrough bleeding events that require hemostatic therapy in addition to Hemlibra prophylaxis
Time Frame: Every 6 months, for the 2 years and 10 months of the patient's study participation duration.
Measure: Number; unit: breakthrough bleeding events
Arm/Group | Single Arm
Number analyzed (Participants) | 1
breakthrough bleeding events | 14

4. Secondary Outcome: Pseudotumor Status
Description: Radiologic evaluation (CT and/or MRI) to evaluate control of progression, stabilization or regression per change in size (measured in cm) of the pseudotumor
Time Frame: Every 12 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient was unable to return for repeat or final assessments of pseudotumor size by radiology scan after baseline assessment due to global COVID19 pandemic. Only baseline measurements were collected and no follow-up measurements, therefore any change in the pseudotumor status could not be evaluated/determined.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Patient Quality of Life Based on Haem-A-QOL
Description: The subjective change in quality of life and activity with Hemlibra (emicizumab) prophylaxis will be evaluated during the study. QoL and activity will be assessed using Haem-A-QoL and EQ-5D-5L. Changes in these measures will be determined by changes from the baseline scores compared to follow-up scores.
Time Frame: Every 12 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient was unable to return for repeat or final QoL assessments after baseline assessment, due to the COVID19 global pandemic. Only baseline measurements were collected and no follow-up measurements, therefore any change in the QoL status could not be evaluated/determined.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Patient Quality of Life Based on EQ-5D-5L
Description: as for outcome 5
Time Frame: Every 12 months, for the 2 years and 10 months of the patient's study participation duration.
Population: as for outcome 5
Arm/Group | Single Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Adverse Events
Description: Number of adverse events while on HemLibra (emicizumab) prophylaxis.
Time Frame: Every 3 months, for the 2 years and 10 months of the patient's study participation duration.
Population: AEs were collected during participant's study participation until study treatment / participation withdrawal.
Measure: Number; unit: adverse events
Arm/Group | Single Arm
Number analyzed (Participants) | 1
adverse events | 3

8. Secondary Outcome: Serious Adverse Events
Description: Number of SAEs while on HemLibra (emicizumab) prophylaxis
Time Frame: Every 3 months, for the 2 years and 10 months of the patient's study participation duration.
Measure: Number; unit: serious adverse events
Arm/Group | Single Arm
Number analyzed (Participants) | 1
serious adverse events | 0

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events while on HemLibra (emicizumab) prophylaxis
Time Frame: Every 3 months, for the 2 years and 10 months of the patient's study participation duration.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 1
participants | 1

10. Secondary Outcome: Anti-Drug Antibodies (ADA)
Description: Development of emicizumab anti-drug antibodies using the ADA assay
Time Frame: Every 12 months, for the 2 years and 10 months of the patient's study participation duration.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 1
participants | 0

11. Secondary Outcome: ADA and Activated Partial Thromboplastin Time (APTT)
Description: If the patient develops an ADA: the ADA's effect on the patient's APTT
Time Frame: Every 12 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient did not develop ADA (anti-drug antibody) during study participation.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

12. Secondary Outcome: ADA and Factor VIII (FVIII)
Description: If the patient develops an ADA: the ADA's effecton the patient's FVIII assay
Time Frame: Every 12 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient did not develop ADA (anti-drug antibody) during study participation.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

13. Secondary Outcome: Planned or Unplanned Surgery
Description: If the patient requires surgery: Whether the procedure(s) was/were planned versus unplanned
Time Frame: Every 6 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient did not require surgery during study treatment.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

14. Secondary Outcome: Hemostatic Agents in Surgery
Description: If the patient requires surgery: Whether hemostatic agents in addition to Hemlibra were required to achieve or maintain hemostasis
Time Frame: Every 6 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient did not require surgery during study participation
Arm/Group | Single Arm
Number analyzed (Participants) | 0

15. Secondary Outcome: Blood Loss in Surgery
Description: If the patient requires surgery: Whether blood loss exceeded the estimated/predicted blood loss relative to a patient without hemophilia
Time Frame: Every 6 months, for the 2 years and 10 months of the patient's study participation duration.
Population: Patient did not have surgery during study participation.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Every 3 months, for the 2 years and 10 months of the patient's study participation duration.
Description: Standard definitions
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=1)
Upper respiratory infection (General disorders) | 1 (1) — Upper respiratory infection
Fall with injurty (Musculoskeletal and connective tissue disorders) | 1 (1)
Malaria infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor wishes to review final study report prior to submission for publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT03921294/Prot_SAP_000.pdf